CLINICAL TRIAL: NCT05125432
Title: Genetic Predictors to Acupuncture Response for Arthralgia Induced by Aromatase Inhibitors in Patients With Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2021006
Record Dates: First submitted 2021-09-27; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Single Nucleotide Polymorphisms; Breast Cancer; Aromatase Inhibitors; Arthralgia; Acupuncture
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture group (Experimental): Acupuncture group Patients with breast cancer who experienced AIA were assessed by the Brief Pain Inventory (BPI)scale and McMasters College Osteoarthritis Index Score (WOMAC). Patients who met the criteria for inclusion would receive regular acupuncture treatment. The location of acupuncture is based on the principles of acupuncture treatment in Traditional Chinese medicine. Patients with high scores and obvious pain received standardized acupuncture treatment, and standard acupuncture points and most painful joint (up to 3) specific point. Meanwhile, blood samples of patients were collected, and SNP related to AIA was screened through SNP typing technology.
  Interventions: Device: Acupuncture group

INTERVENTIONS:
Device: Acupuncture group — Acupuncture group Patients with breast cancer who experienced AIA were assessed by the Brief Pain Inventory (BPI)scale and McMasters College Osteoarthritis Index Score (WOMAC). Patients who met the criteria for inclusion would receive regular acupuncture treatment. The location of acupuncture is based on the principles of acupuncture treatment in Traditional Chinese medicine. Patients with high scores and obvious pain received standardized acupuncture treatment, and standard acupuncture points and most painful joint (up to 3) specific point. Meanwhile, blood samples of patients were collected, and SNP related to AIA was screened through SNP typing technology.

SUMMARY:
Purpose:Acupuncture for arthralgia induced by aromatase inhibitors in patients with breast cancer associated with screening of SNPs.

DETAILED DESCRIPTION:
Aromatase inhibitor-induced arthralgia (AIA) is the most common side effect of aromatase inhibitors (AIs) used in breast cancer , may cause poor adherence to AIs. Studies have shown that acupuncture has a certain therapeutic effect on AIA in breast cancer. In this study, acupuncture was used to relieve the symptoms of arthralgia in patients, and the efficacy of acupuncture was observed by using relevant scales. Currently, studies have shown that AIA in breast cancer patients is related to some biological factors.

At the same time, we collected peripheral blood samples of patients, combined with the reported relevant literature, screened out the single nucleotide polymorphisms(SNP) related to AIA and to guide acupuncture treatment of aromatase Inhibitors induced arthralgia, balance the toxicity of endocrine therapy, and improve compliance and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. History of stage I-III breast cancer and free of disease by clinical examination;Currently receiving aromatase inhibitors (Anastrozole, Letrozole, or Exemestane) treatment;
2. AI-assisted treatment has lasted for more than one month, and there are obvious symptoms of arthralgia ;
3. Voluntarily participate in the clinical trial and sign the informed consent form after informed consent (patients voluntarily accept the treatment and give informed consent);
4. Eastern Cooperative Oncology Group (ECOG) score of physical condition (0-1);
5. Patients with previous local recurrence were eligible, but not patients with distant metastasis;
6. The basic indexes were consistent, and the blood routine and ECG were normal.

Exclusion Criteria:

1. Patients with needle phobia;
2. Low platelet count (<50000); comorbidity with a bleeding disorder; comorbidity with thyroid dysfunction; pregnancy; haemoglobin levels <10 g/dl and haematocrit <30; anaemia on active pharmacological treatment orreceiving blood transfusion or steroids;
3. Lymphoedematous of limbs;
4. Patients have a history of acupuncture treatment for 6 months;
5. Patients were reluctant to participate in the study;
6. A prior history of inflammation, metabolic disease, or neurotic joints, except for previous treatment with bisphosphonates, steroids, or opioid analgesics.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2021-11-25 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in arthralgia scores were measured by the BPI | 52 weeks
  Changes in arthralgia scores were measured by the Brief Pain Inventory (BPI) before and after acupuncture treatment.

SECONDARY OUTCOMES:
Changes in arthralgia scores were measured by the WOMAC scales | 52 weeks
  Changes in arthralgia scores were measured by the McMasters College Osteoarthritis Index Score (WOMAC) scales before and after acupuncture treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qinghai University, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: No